CLINICAL TRIAL: NCT01396941
Title: Effects of Sleep Duration and Architecture on Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K23HL096832 (NIH); K23HL096832 (NIH)
Record Dates: First submitted 2011-07-15; First posted 2011-07-19 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Insulin Resistance
Keywords: Diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sleep restriction (Experimental): The investigators will compare the effects of sleep restriction vs. normal sleep in healthy volunteers, using a randomized crossover study design. Each subject will undergo a period of normal sleep and a period of sleep restriction, separated by a 1-month washout period. Subjects will be randomized to receive either sleep restriction first (later followed by normal sleep) or normal sleep first (later followed by sleep restriction).
  Interventions: Behavioral: Sleep restriction

INTERVENTIONS:
Behavioral: Sleep restriction — Sleep restriction will consist of 5 nights, sleeping 4 hours per night Normal sleep will consist of 5 nights, sleeping 9 hours per night

SUMMARY:
This pilot clinical trial will test the hypotheses that sleep restriction (for 5 nights), in comparison to "normal sleep", will:

1. Decrease peripheral insulin sensitivity and glucose tolerance, as measured by the hyperinsulinemic-euglycemic clamp and oral glucose tolerance test.
2. Decrease hepatic insulin sensitivity, as assessed by stable isotope studies of endogenous glucose production, gluconeogenesis and glycogenolysis.

DETAILED DESCRIPTION:
Over the past 50 years, the incidence of diabetes has increased dramatically, while sleep duration in the US has decreased significantly. Epidemiological studies and small clinical trials suggest that these trends are causally related. In this study, our goal is to determine the mechanisms by which decreased sleep duration directly affects insulin sensitivity. The investigators will perform a clinical study in 20 healthy volunteers to determine whether 5 nights of sleep restriction decreases insulin sensitivity in the peripheral tissues (ie, skeletal muscle) or liver.

Peripheral insulin sensitivity will be measured by the hyperinsulinemic-euglycemic clamp, and hepatic insulin sensitivity will be quantified by measurement of hepatic glucose production, gluconeogenesis and glycogenolysis (using stable isotope tracer methods). Subjects will be randomized to an initial period of "normal sleep" or sleep restriction and will be admitted to the Clinical Research Center (CRC) for 9 days to undergo comprehensive metabolic studies and sleep assessments under the assigned sleep condition. After a 1-month washout period, subjects will be re-admitted to the CRC to undergo these same assessments under the opposite sleep condition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Regular work hours (ie, no night-time or shift work within the past 6 months)
* Pittsburgh Sleep Quality Index (PSQI) Score <5
* Average nightly sleep duration 6-9 hours (per screening actigraphy)

Exclusion Criteria:

* Current or prior diabetes, gestational diabetes, impaired glucose tolerance or impaired fasting glucose
* Type 2 diabetes in biological parents
* BMI >=25
* Pregnancy
* Chronic medical condition, including: psychiatric disorders, heart disease, pulmonary disease, infectious diseases, rheumatological and neurological disorders
* Use of prescribed medications on a regular basis.
* History of disorder involving hypothalamic, pituitary or adrenal glands
* History of or current sleep disorders (insomnia, restless leg syndrome, sleep disordered breathing, narcolepsy, etc)
* Anemia
* Cognitive impairment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 1 month
  Peripheral insulin sensitivity will be measured using the hyperinsulinemic-euglycemic clamp. Hepatic insulin sensitivity will be measured using stable isotope tracer studies.

CONTACTS AND LOCATIONS:
Overall Officials: Madhu N. Rao, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF San Francisco General Hospital, San Francisco, California, United States